CLINICAL TRIAL: NCT03170713
Title: Impact of Preemptive Intravenous Ibuprofen on Postoperative Edema and Trismus in the Third Molar Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, assist. prof., Erzincan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ERZINCAN UNIVERSITY 10
Record Dates: First submitted 2017-05-20; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Trismus; Edema
Keywords: Preemptive intravenous ibuprofen; trismus; edema; Third molar tooth extraction; Antiinflammatory effect
MeSH Terms: conditions — Trismus; Edema | interventions — dexketoprofen trometamol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- arveles (Active Comparator): 800 mg ibuprofen and 50 mg arveles in 150 cc normal saline before operation will be given in 30 minutes.
  Interventions: Drug: arveles; Drug: intrafen; Other: placebos
- intrafen (Active Comparator): intrafen 800 mg in 150 cc normal saline before operation will be given in 30 minutes.
  Interventions: Drug: arveles; Drug: intrafen; Other: placebos
- placebos (Placebo Comparator): Pre-operative 150 cc normal saline will be delivered in 30 minutes
  Interventions: Drug: arveles; Drug: intrafen

INTERVENTIONS:
Drug: arveles — 800 mg ibuprofen and 50 mg dexketoprofen in 150 cc normal saline before operation will be given in 30 minutes. The edema size, mouth opening (trismus) will be recorded in all patients in the preoperative period, postoperative period, postoperative 48th hour and 1 st week.
  Other Names: dexketoprofen
Drug: intrafen — 800 mg ibuprofen in 150 cc normal saline before operation will be given in 30 minutes.The edema size, mouth opening (trismus) will be recorded in all patients in the preoperative period, postoperative period, postoperative 48th hour and 1 st week.
  Other Names: ibuprofen i.v.
Other: placebos — 150 cc normal saline before operation will be given in 30 minutes.The edema size, mouth opening (trismus) will be recorded in all patients in the preoperative period, postoperative period, postoperative 48th hour and 1 st week.
  Arms: arveles; intrafen

SUMMARY:
this study was planned to investigate the antiinflammatory activity of preemptive intravenous ibuprofen on inflammatory complications such as edema and trismus after third molar tooth surgery

ELIGIBILITY:
Inclusion Criteria:

* Elective 3. Molar tooth extraction
* Patients between the ages of 20-35
* Patients who are symptomatic
* 3. Molar tooth angular or horizontal settled patients

Exclusion Criteria:

* Patients who refuse to participate in the study
* Patients under 20 years old, over 35 years old
* Patients who are allergic to known non-steroidal anti-inflammatory drugs
* Pregnant patients
* Patients with severe hepatic insufficiency
* Patients with severe renal insufficiency

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-10-30 (Estimated); Study Completion 2017-11-15 (Estimated)

PRIMARY OUTCOMES:
Edema size measured by tape measure method | 6 month
  the effect of preemptive intravenous ibuprofen on postoperative edema size

SECONDARY OUTCOMES:
Maximum mouth opening measured with vernier caliper | 6 month
  the effect of preemptive intravenous ibuprofen on postoperative trismus rate

CONTACTS AND LOCATIONS:
Overall Officials: ilke kupeli, Principal Investigator — Erzincan University
Locations (1):
- Erzincan University, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jerjes W, El-Maaytah M, Swinson B, Banu B, Upile T, D'Sa S, Al-Khawalde M, Chaib B, Hopper C. Experience versus complication rate in third molar surgery. Head Face Med. 2006 May 25;2:14. doi: 10.1186/1746-160X-2-14. PMID 16725024
- [Background] Bouloux GF, Steed MB, Perciaccante VJ. Complications of third molar surgery. Oral Maxillofac Surg Clin North Am. 2007 Feb;19(1):117-28, vii. doi: 10.1016/j.coms.2006.11.013. PMID 18088870
- [Background] Chukwuneke F, Onyejiaka N. Management of postoperative morbidity after third molar surgery: a review of the literature. Niger J Med. 2007 Apr-Jun;16(2):107-12. doi: 10.4314/njm.v16i2.37291. PMID 17694761
- [Background] Colorado-Bonnin M, Valmaseda-Castellon E, Berini-Aytes L, Gay-Escoda C. Quality of life following lower third molar removal. Int J Oral Maxillofac Surg. 2006 Apr;35(4):343-7. doi: 10.1016/j.ijom.2005.08.008. Epub 2005 Nov 8. PMID 16280233
- [Background] Vegas-Bustamante E, Mico-Llorens J, Gargallo-Albiol J, Satorres-Nieto M, Berini-Aytes L, Gay-Escoda C. Efficacy of methylprednisolone injected into the masseter muscle following the surgical extraction of impacted lower third molars. Int J Oral Maxillofac Surg. 2008 Mar;37(3):260-3. doi: 10.1016/j.ijom.2007.07.018. Epub 2008 Mar 4. PMID 18296027
- [Background] Chukwuneke FN, Oji C, Saheeb DB. A comparative study of the effect of using a rubber drain on postoperative discomfort following lower third molar surgery. Int J Oral Maxillofac Surg. 2008 Apr;37(4):341-4. doi: 10.1016/j.ijom.2007.11.016. Epub 2008 Feb 12. PMID 18272338
- [Result] Sato FR, Asprino L, de Araujo DE, de Moraes M. Short-term outcome of postoperative patient recovery perception after surgical removal of third molars. J Oral Maxillofac Surg. 2009 May;67(5):1083-91. doi: 10.1016/j.joms.2008.09.032. PMID 19375022
- [Result] Markovic A, Todorovic Lj. Effectiveness of dexamethasone and low-power laser in minimizing oedema after third molar surgery: a clinical trial. Int J Oral Maxillofac Surg. 2007 Mar;36(3):226-9. doi: 10.1016/j.ijom.2006.10.006. Epub 2006 Dec 8. PMID 17157479
- [Result] Jain N, Maria A. Randomized double blind comparative study on the efficacy of Ibuprofen and aceclofenac in controlling post-operative sequelae after third molar surgery. J Maxillofac Oral Surg. 2011 Jun;10(2):118-22. doi: 10.1007/s12663-011-0198-9. Epub 2011 Apr 22. PMID 22654361
- [Result] Agarwal S, Chattopadhyay S, Mandal M. Comparison of efficacy of aceclofenac and ibuprofen after surgical removal of impacted third molar. J. Evolution Med. Dent. Sci. 2017;6(21):1670-1677, DOI: 10.14260/Jemds/2017/368